CLINICAL TRIAL: NCT00126997
Title: Blinded, Randomised Study to Assess the Immunogenicity and Safety of GlaxoSmithKline (GSK) Biologicals' Live Attenuated Measles-mumps-rubella-varicella Candidate Vaccine When Given to Healthy Children in Their Second Year of Life
Brief Title: Immunogenicity and Safety of Combined Vaccine to Prevent Measles, Mumps, Rubella and Chickenpox Diseases
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 104020
Record Dates: First submitted 2005-08-04; First posted 2005-08-05 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Mumps; Rubella; Measles; Varicella
Keywords: Prophylaxis measles, mumps, rubella and chickenpox
MeSH Terms: conditions — Mumps; Rubella; Measles; Chickenpox | interventions — Vaccines, Attenuated

INTERVENTIONS:
Biological: Measles, Mumps, Rubella and Chickenpox (live vaccine)

SUMMARY:
This is a study to assess the immunogenicity and safety of GlaxoSmithKline (GSK) Biologicals live attenuated measles-mumps-rubella-varicella vaccine given to healthy children in their second year of life.

ELIGIBILITY:
Inclusion Criteria:

* A male or female subject between 11-13 months of age (i.e. from 11 month birthday until the day before the 14 month birthday) at the time of the first vaccination.

Exclusion Criteria:

* History of previous measles, mumps, rubella and/or varicella vaccination or disease, or known exposure to any of these diseases within 30 days prior to the start of the trial
* Planned administration of a vaccine not foreseen by the study protocol from 30 days prior to each vaccination until 42-56 days after each vaccination

Ages: 11 Months to 21 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1439 (Actual)
Dates: Start 2005-05; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Antibody levels after vaccination.

SECONDARY OUTCOMES:
Safety of the study vaccines.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (52):
- Finland (7):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Lahti
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
  - GSK Investigational Site, Vantaa
- Germany (35):
  - GSK Investigational Site, Bayreuth, Bavaria
  - GSK Investigational Site, Bindlach, Bavaria
  - GSK Investigational Site, Bobingen, Bavaria
  - GSK Investigational Site, Cham, Bavaria
  - GSK Investigational Site, Kempten (Allgäu), Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nördlingen, Bavaria
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Olching, Bavaria
  - GSK Investigational Site, Tegernsee, Bavaria
  - GSK Investigational Site, Tutzing, Bavaria
  - GSK Investigational Site, Veitshöchheim, Bavaria
  - GSK Investigational Site, Eschwege, Hesse
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Fulda, Hesse
  - GSK Investigational Site, Nidderau, Hesse
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Salzgitter, Lower Saxony
  - GSK Investigational Site, Wolfenbüttel, Lower Saxony
  - GSK Investigational Site, Bad Oeynhausen, North Rhine-Westphalia
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Detmold, North Rhine-Westphalia
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Espelkamp, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Gütersloh, North Rhine-Westphalia
  - GSK Investigational Site, Hille, North Rhine-Westphalia
  - GSK Investigational Site, Kirchlengern, North Rhine-Westphalia
  - GSK Investigational Site, Krefeld, North Rhine-Westphalia
  - GSK Investigational Site, Löhne, North Rhine-Westphalia
  - GSK Investigational Site, Minden, North Rhine-Westphalia
  - GSK Investigational Site, Mönchengladbach, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Wesseling, North Rhine-Westphalia
  - GSK Investigational Site, Willich, North Rhine-Westphalia
- Greece (5):
  - GSK Investigational Site, Arta
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Komotini
  - GSK Investigational Site, Rhodes
  - GSK Investigational Site, Thessaloniki
- Poland (5):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Siemianowice Śląskie
  - GSK Investigational Site, Trzebnica

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 104020 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104020 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104020 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104020 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104020 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104020 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register